CLINICAL TRIAL: NCT05636553
Title: Mixed-methods Single-arm Study Evaluating the Feasibility of Massage as an Adjunct Approach to Care for Pregnant Women Who Have Experienced a Stillbirth
Brief Title: Massage as an Adjunct Approach to Care for Pregnant Women Who Have Experienced a Stillbirth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fogarty Sarah (Other)
Collaborators: Massage Therapy Foundation (Other); University of Western Sydney (Other)
Responsible Party: Principal Investigator, Sarah Fogarty, Principal Investigator, Fogarty Sarah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20705.66430
Record Dates: First submitted 2022-11-11; First posted 2022-12-05 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Pregnancy Related; Pregnancy Loss
Keywords: pregnancy; massage; pregnancy after stillbirth
MeSH Terms: interventions — Massage

STUDY DESIGN:
Intervention Model Description: A convergent parallel mixed-methods, single arm repeated measures pilot trial design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Massage (Experimental): Women will receive four 60 minute massage consultations within a four-month period at intervals of their choosing.
  Interventions: Other: Massage

INTERVENTIONS:
Other: Massage — Individualised treatment using massage techniques such as longitudinal gliding, transverse gliding, digital ischemic pressure, transverse frictions, and transverse gliding.

SUMMARY:
The goal of this mixed-methods single-arm study is to measure the feasibility of massage as an adjunct approach to care for pregnant women who have experienced a stillbirth. In order to provide pilot data, this intervention study will:

1. Determine the feasibility and acceptability of the massage intervention and optimize the timing and outcome measures,
2. Provide data for future use in an individual participant data systematic review, and
3. Evaluate experiences of women undertaking the intervention

Participants will [ If there is a comparison group: Researchers will compare [insert groups] to see if [insert effects].

DETAILED DESCRIPTION:
Research shows that women experiencing pregnancy after stillbirth experience anxiety, fear, and depression. There is a limited evidence of adjunct emotional care approaches for women to utilise to help manage pregnancy after a stillbirth. Massage may assist women who are pregnant after a stillbirth via decreasing anxiety, worry and stress.

Aim: To measure the feasibility of massage as an adjunct approach to care for pregnant women who have experienced a stillbirth.

Design: This study will use a convergent parallel mixed-methods, single arm repeated measures pilot trial design.

Setting: Massage therapists' private clinics across Australia. Participants: Subjects will include 75 pregnant women who have experienced a stillbirth in a previous pregnancy.

Intervention: Women will receive four massages within a four-month period at intervals of their choosing. The massage treatments are based on a vulnerability-to-stress concept which acknowledges the impact of stress on a pregnant woman based on a biopsychosocial model.

The massage protocol allows treatment to be individualised to meet the needs of the participant.

Main outcome measures: The primary outcomes are a) feasibility, b) acceptability and experience of the massage intervention and c) optimization - i.e., capacity of the outcome measures to capture the impact of the intervention received, and to determine when treatments are likely to be of most value.

Analysis Plan: Data will be analysed to meet the study objectives of determining feasibility, acceptability, optimising timing, and outcome measures, and to obtain preliminary data to understand the effects and value of massage on women who are pregnant after a stillbirth.

Significance of the work: Standard antenatal care is emotionally unsuitable for many women in pregnancies following a stillbirth and there is a lack of direct evidence on what interventions or approaches to care might benefit these women. Our proposed research will begin to address this lack of direct evidence.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women 18 years of age or greater who have experienced a stillbirth (pregnancy loss from 20 weeks gestation) in a previous pregnancy.
* Participants who had a medial termination from 20-weeks' gestation will be included in the study.
* Participants must be able to attend one of the study pregnancy massage therapists' clinics located within Australia.
* Having had previous massage experience is not an enrolment criterion, it is just not an exclusion criterion.

Exclusion Criteria:

- Participants will be excluded if they are unable to receive the study treatments in the allocated time frame.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
To assess the feasibility of massage as an adjunct approach to care for pregnant women who have experienced a stillbirth as assessed using a mixed methods narrative and joint display approach | 1 year
  The quantitative and qualitative findings will be integrated using a narrative reporting approach and fit of data integration (coherence of the quantitative and qualitative findings) will be reported.

SECONDARY OUTCOMES:
Changes in worry from baseline to a week post treatment interventions using the self-reported Cambridge Worry Score | Through study completion, an average of 1 year
  Higher scores indicate greater worry. Scores from 0-85
Changes in maternal anxiety symptoms from baseline to a week post treatment interventions using the Generalized Anxiety Disorder Assessment 7 | Through study completion, an average of 1 year
  Higher scores indicate greater anxiety. Min score is 0 and max is 21.
Changes in coping from baseline to a week post treatment interventions using the self-reported Revised Prenatal Coping Inventory | Through study completion, an average of 1 year
  Higher scale scores correspond to a more frequent use of the specific coping style.
Changes in self-efficacy from baseline to a week post treatment interventions using the Strategies Used by People to Promote Health measure | Through study completion, an average of 1 year
  Higher scores indicate greater confidence in carrying out the behaviors to promote health. Total score range is from 29 to 145.
Changes in maternal stress symptoms from baseline to a week post treatment interventions using the Perceived Stress Scale | Through study completion, an average of 1 year
  Higher scores indicating higher perceived stress. The total score range is from zero to 40 with a scores ranging from 0-13 considered low stress, 14-26 moderate stress and 27-40 high stress.
Assessing empathy in the context of the therapeutic relationship via the Consultation and Relational Empathy patient-reported experience measure | Through study completion, an average of 1 year
  This scale has 10 items that measures patients' perceptions of relational empathy in the consultation. The total score range is from 10 to 40 with higher scores indicating greater perceived relational empathy.
Recruitment rates (proportion of people randomised/proportion of people eligible) | Through study completion, an average of 1 year
  Presented as numbers and percentages
Retention rates (proportion of people providing the outcomes of interest/proportion randomised) | Through study completion, an average of 1 year
  Presented as numbers and percentages
Compliance with completing the validated outcome measures (number of validated measures asked to complete/number of validated measures completed) | Through study completion, an average of 1 year
  Presented as numbers and percentages
Elucidating participants' experience of massage in a pregnancy after a stillbirth using a qualitative in-depth interview | Through study completion, an average of 1 year
  Thematic inductive analysis will be used to analyse the qualitative data
Optimization of massage timing to determine when treatments are likely to be of most value presented as a average of time between treatments | Through study completion, an average of 1 year
  Presented as means and ranges of times between treatments

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Fogarty, PhD, Principal Investigator — Western Sydney University
Locations (1):
- Western Sydney University, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in a publication. The stored data available for re-use will not have information in it that makes participants identifiable.
Time Frame: Data collected from this study will be made available online and world-wide in perpetuity.
Access Criteria: None, it will be open access.
URL: https://researchdirect.westernsydney.edu.au